CLINICAL TRIAL: NCT02766751
Title: Treating Comorbid Pain and Depression in HIV+ Individuals
Acronym: HIVPass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Responsible Party: Principal Investigator, Michael Stein, MD, Principal Investigator, Butler Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 840019
Record Dates: First submitted 2016-05-06; First posted 2016-05-10 (Estimated); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: HIV; Depression; Pain
MeSH Terms: conditions — Depression; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health Education (Placebo Comparator): The seven sessions will cover: 1) nutrition (2 sessions), 2) sleep hygiene, 3) building immunity (e.g., how to avoid colds/flu), 4) injury/disease prevention (e.g., seat belts, sunscreen, when to get regular check-ups/screenings etc.), 5) benefits of exercise/cardiac health, 6) alternative medicine (massage, acupuncture). These sessions will be primarily didactic and consist of health education, followed by discussion as to how this information compares to that which the participants may have been exposed to in the past.
  Interventions: Behavioral: Health Education
- HIVPASS (Experimental): Over 7 sessions, the interventionist and the participant will explore the relationship between pain, depressive symptoms, and HIV. General information about pain, HIV and depression will be discussed, as will avoidance of physical activity. Psychoeducation about these areas will be tied to the participant's stated life goals, and exposure exercises and goal lists will be developed. Later sessions will integrate continued efforts towards reaching goals and reducing avoidance. A release of information will be obtained from the participant to allow study session chart notes to be placed in the medical record at the participant's PCP office and to allow the PCP and the study interventionist to discuss treatment coordination.
  Interventions: Behavioral: HIVPASS

INTERVENTIONS:
Behavioral: HIVPASS — The 7-session HIVPASS intervention is provided to individuals randomized to the HIVPASS study arm.
  Arms: HIVPASS
Behavioral: Health Education — The 7-sessions of Health Education is provided to individuals randomized to the Health Education study arm.
  Arms: Health Education

SUMMARY:
This study is designed to look at two different programs that may help people who are HIV+ and have pain and depression. The investigators are trying to understand how to help people learn to live better lives even with these chronic illnesses.

DETAILED DESCRIPTION:
The primary aim of this RCT is to evaluate the HIVPass intervention. HIV+ participants (n=236) with chronic pain and depression will be recruited at primary care HIV Clinics through posted advertisements in the waiting rooms of the PCP offices and by physician referral. After an initial phone study screen, research staff will meet with interested individuals in their PCP offices for informed consent, baseline interview and randomization into one of two study groups (Health Education or HIVPass Counseling). Seven intervention sessions (HE or HIVPASS) will occur during the first 3 months of study participation. For all participants, the first session is a collaborative in-person joint session with the participant, his/her PCP and the study BHS. Session 2 is conducted immediately after this collaborative session, and is also in-person. Sessions 3-7 are conducted by phone. Follow-up assessment interviews will be at months 1, 2, 3 (post-intervention), 4, 6, 9 and 12.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Pain (pain duration for at least six months with a mean score of greater than 3.5 on the BPI Pain Interference Scale)
* Pain severity > or equal to 4 on a Numeric Rating Scale indicating "average pain in the last week"
* At least one trial of PCP-recommended medication (i.e. acetaminophen, NSAIDS, muscle relaxants) judged through interviews with patients and PCPs
* Quick Inventory of Depression Symptoms (QIDS) score of ≥ 9 (depression severity)
* Stable dose of an antidepressant, if using, for the previous 1 months
* Age > or equal to 18
* HIV+
* Planning to live in the area for the next 6 months
* Access to a telephone that is typically working.

Exclusion Criteria:

* In psychotherapy or a multidisciplinary pain management program
* Planned surgery in the next 6 months
* Pain thought due to cancer
* Current mania
* Past year chronic psychotic condition
* Excessive substance use (Use of cocaine, heroin, or non-prescribe opioids 15 days per month or more; binge alcohol use 4 days per month or more)
* Suicidality requiring immediate attention
* Pregnancy or planned pregnancy in the next 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
pain interference | 3 months
  Brief pain inventory, interference scale

SECONDARY OUTCOMES:
depression | 3 months; 12 months
  Quick Inventory of depression symptoms
activity level | 3 months; 12 months
  Assessed with actigraphy
anxiety | 3 months; 12 months
  State-Trait Anxiety Inventory
viral load | 3 months, 12 months
ART adherence | 3 months, 12 months
  AIDS Clinical Trial Group questionnaire
perception of global improvement | 3 months, 12 months
  Patient Global Impression of Change Scale
health related quality of life | 3 months, 12 onths
  Short Form 36 Health Survey
pain interference | 12 months
  brief pain inventory, interference scale

CONTACTS AND LOCATIONS:
Overall Officials: Michael Stein, MD, Principal Investigator — Butler Hospital
Locations (4):
- United States (4):
  - Boston University/Boston Medical Center, Boston, Massachusetts
  - Hennepin Healthcare, Minneapolis, Minnesota
  - Butler Hospital, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Uebelacker LA, Pinkston MM, Busch AM, Baker JV, Anderson B, Caviness CM, Herman DS, Weisberg RB, Abrantes AM, Stein MD. HIV-PASS (Pain and Sadness Support): Randomized Controlled Trial of a Behavioral Health Intervention for Interference Due to Pain in People Living With HIV, Chronic Pain, and Depression. Psychosom Med. 2023 Apr 1;85(3):250-259. doi: 10.1097/PSY.0000000000001172. Epub 2023 Feb 3. PMID 36799731
- [Derived] Pinkston MM, Busch AM, Stein M, Baker J, Caviness C, Herman D, Weisberg R, Abrantes AM, Uebelacker LA. Improving functioning in HIV+ patients with chronic pain and comorbid depression: Protocol for a randomized clinical trial testing a collaborative behavioral health intervention based on behavioral activation. Contemp Clin Trials. 2022 Aug;119:106842. doi: 10.1016/j.cct.2022.106842. Epub 2022 Jun 28. PMID 35777696